CLINICAL TRIAL: NCT04745884
Title: Early Non-invasive Detection of Progression of Mass Effect From Unilateral Brain Lesions
Brief Title: A Study to Detect Progression of Mass Effect From Unilateral Brain Lesions
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Device sensitive issues
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Alejandro Rabinstein, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 20-009516
Record Dates: First submitted 2021-02-04; First posted 2021-02-09 (Actual); Results first posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-12

CONDITIONS: Non-traumatic Hemispheric Brain Lesions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Monitoring (Experimental): Imaging guided by monitoring results
  Interventions: Device: Non-invasive bilateral monitoring of ICP waveform

INTERVENTIONS:
Device: Non-invasive bilateral monitoring of ICP waveform — Brain4care non-invasive bilateral monitoring of ICP waveform

SUMMARY:
The purpose of this research is to gather information on the safety and effectiveness of the Brain4Care device for measuring intracranial pressure without invasive procedures.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with non-traumatic hemispheric brain lesions deemed at risk for progression of mass effect and possible subfalcine and/or uncal herniation.
* Patients admitted the Neuroscience ICU for serial neurological monitoring.
* Patients whose care is not expected to include immediate surgical decompression.

Exclusion Criteria:

* Patients under the age of 18.
* Patients who are unable to provide consent due to neurologic deficit and does not have a surrogate decision maker available to provide consent.
* Known or suspected Pregnancy
* Adults with cranial defects or that have undergone craniectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-02-04 (Actual); Primary Completion 2024-12-02 (Actual); Study Completion 2024-12-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Rabinstein, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment stopped because bilateral monitoring was proven not sufficiently reliable for investigation
Period: Overall Study
Arm/Group | Monitoring
Started | 6
Completed | 3
Not Completed | 3
Not completed — Excessive Signal Feedback-Uninterpretable Data | 3

BASELINE CHARACTERISTICS:
Arm/Group | Monitoring
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Functional Outcome
Description: Functional outcome was assessed using the Modified Rankin Scale (mRS) which assesses functional outcomes in patients recovering from strokes. It consists of a 7-point ordinal scale ranging from 0 to 6 where 0=no symptoms and 6=dead with higher scores indicating a worse functional outcome.
Time Frame: 3 months
Population: 1 patient was unable to be reached for follow up
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | Monitoring
Number analyzed (Participants) | 5
score on a scale | 3 [2 to 4]

2. Secondary Outcome: Imaging Utilization
Description: Number of imaging scans
Time Frame: within ICU admission
Population: The BrainCare device was too sensitive to any movement including breathing. Due to the sensitivity of the device, zero ICP waveforms were detected. The waveforms were needed to measure this outcome, with the waveforms not showing up on the BrainCare device due to the sensitivity of the device, this outcome could not be measured.
Arm/Group | Monitoring
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of informed consent through study completion, approximately 3 months.
Arm/Group | Monitoring
All-Cause Mortality (participants affected / at risk) | 2/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

LIMITATIONS AND CAVEATS:
The study was terminated early as there were issues with the sensitive of the device.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2021-01-06): https://cdn.clinicaltrials.gov/large-docs/84/NCT04745884/Prot_000.pdf